CLINICAL TRIAL: NCT04847479
Title: Close Contact Self-Testing Among Contacts of Individuals With COVID-19 Infection
Brief Title: COVID-19 Close Contact Self-Testing Study
Acronym: CloseST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Public Health Management Corporation (Other)
Responsible Party: Principal Investigator, Robert Gross, Professor of Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3R01HL151292-01S1-2; 3R01HL151292-01S1 (NIH)
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Test kit distribution (Experimental): Participants in the self-test arm receive multiple COVID-19 self-test kits to distribute to their close contacts.
  Interventions: Behavioral: COVID-19 self-test
- Test referral distribution (Active Comparator): Participants in the test referral arm receive text messages providing testing information to send to their close contacts.
  Interventions: Behavioral: COVID-19 test referral

INTERVENTIONS:
Behavioral: COVID-19 self-test — Up to 3 COVID-19 self-test kits will be given to individuals who have tested positive for COVID-19. Participants will be instructed to give test kits to close contacts who have been exposed to them.
  Arms: Self-Test kit distribution
Behavioral: COVID-19 test referral — Text messages with testing information will be given to individuals who have tested positive for COVID-19. Participants will be instructed to share text messages with close contacts who have been exposed to them.
  Arms: Test referral distribution

SUMMARY:
Widespread testing and contact tracing are critical to controlling the COVID-19 epidemic. Distribution of COVID-19 self-test kits can augment public health contact tracing efforts, as individuals with COVID-19 can distribute self-testing to close contacts. This approach can increase case detection by facilitating testing among exposed individuals, and potentially ameliorate stigma, fear, and medical mistrust associated with COVID-19 among vulnerable populations.

The central hypothesis of this study is that distribution of SARS-CoV-2 self-tests to close contacts of among individuals with COVID-19 infection can increase case detection compared with a standard contact referral strategy.

DETAILED DESCRIPTION:
Strategies to increase testing among individuals exposed to COVID-19 are needed. One approach to increase testing and case detection is to distribute home test kits to close contacts of individuals with COVID-19. This approach decreases logistic barriers to testing, potential exposures to COVID-19, and reduces potential stigma and fear associated with facility-based COVID-19 testing.

The investigators will conduct a cohort study of individuals diagnosed with COVID-19 in the C-STRAND trial (NCT04797858), in order to determine if distribution of self-test kits to close contacts of of individuals with COVID-19 can increase case detection compared with a standard contact referral strategy among. Individuals diagnosed with COVID-19 who were randomized to the self-test (intervention) arm or received self-test kits will be assigned to receive additional self-test kits to distribute to close contacts. Individuals diagnosed with COVID-19 who were randomized to the test referral (control) arm or received test referrals will be assigned to receive text message referrals to give their close contacts to seek testing if needed. COVID-19 case detection and test uptake will be measured in both arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has a working telephone number
* Willing and able to provide informed consent

Exclusion Criteria:

* Severe symptoms requiring immediate medical attention
* Younger than 18 years of age
* Does not have a working telephone number
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gross, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Public Health Management Corporation, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bien-Gund C, Dugosh K, Acri T, Brady K, Thirumurthy H, Fishman J, Gross R. Factors Associated With US Public Motivation to Use and Distribute COVID-19 Self-tests. JAMA Netw Open. 2021 Jan 4;4(1):e2034001. doi: 10.1001/jamanetworkopen.2020.34001. PMID 33471114
- [Background] Lightfoot MA, Campbell CK, Moss N, Treves-Kagan S, Agnew E, Kang Dufour MS, Scott H, Sa'id AM, Lippman SA. Using a Social Network Strategy to Distribute HIV Self-Test Kits to African American and Latino MSM. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):38-45. doi: 10.1097/QAI.0000000000001726. PMID 29771792
- [Background] Thirumurthy H, Masters SH, Mavedzenge SN, Maman S, Omanga E, Agot K. Promoting male partner HIV testing and safer sexual decision making through secondary distribution of self-tests by HIV-negative female sex workers and women receiving antenatal and post-partum care in Kenya: a cohort study. Lancet HIV. 2016 Jun;3(6):e266-74. doi: 10.1016/S2352-3018(16)00041-2. Epub 2016 Apr 8. PMID 27240789
- [Background] Altamirano J, Govindarajan P, Blomkalns AL, Kushner LE, Stevens BA, Pinsky BA, Maldonado Y. Assessment of Sensitivity and Specificity of Patient-Collected Lower Nasal Specimens for Severe Acute Respiratory Syndrome Coronavirus 2Testing. JAMA Netw Open. 2020 Jun 1;3(6):e2012005. doi: 10.1001/jamanetworkopen.2020.12005. PMID 32530469
- See also: C-STRAND Trial — https://clinicaltrials.gov/ct2/show/NCT04797858

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We were unable to recruit participants in the test referral distribution arm since there were no patients in that arm that tested positive.
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [26 to 42] |  | 33 [26 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 2 |  | 2
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Positive Contacts
Description: Number of close contacts who test positive for COVID-19
Time Frame: 8 weeks
Population: We were unable to recruit any participants in the test referral arm who tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 3 | 0
Participants | 0 | 0

2. Secondary Outcome: Number of Positive Contacts (End of Study)
Description: Number of close contacts who test positive for COVID-19 by the end of the study
Time Frame: Through study completion, up to one year
Population: We were unable to recruit any participants in the test referral arm who tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 3 | 0
Participants | 0 | 0

3. Secondary Outcome: Number of Contacts Tested
Description: Number of close contacts who completed a test
Time Frame: 8 weeks
Population: We were unable to recruit any participants in the test referral arm who tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 3 | 0
Participants | 2 |

4. Secondary Outcome: Number of Contacts Tested (End of Study)
Description: Number of close contacts who completed a test by the end of the study
Time Frame: Through study completion, up to one year
Population: We were unable to recruit any participants in the test referral arm who tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 3 | 0
Participants | 0 | 0

5. Secondary Outcome: Number of Household Contacts Tested
Description: Number of household contacts who completed a test
Time Frame: 8 weeks
Population: We were unable to recruit any participants in the test referral arm who tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 3 | 0
Participants | 0 | 0

6. Secondary Outcome: Number of Household Contacts Tested (End of Study)
Description: Number of household contacts who completed a test by the end of the study
Time Frame: Through study completion, up to one year
Population: We were unable to recruit any participants in the test referral arm who tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 3 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were considered enrolled in our study for 8 weeks. 8 weeks after enrollment, they completed a follow-up survey and were then considered to have completed the study.
Description: We were unable to recruit any participants in the test referral arm who tested positive.
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT04847479/Prot_SAP_000.pdf